CLINICAL TRIAL: NCT00598572
Title: Safety and Tolerability of Deferoxamine in Acute Cerebral Hemorrhage
Brief Title: Dose Finding and Safety Study of Deferoxamine in Patients With Brain Hemorrhage
Acronym: DFO In ICH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Massachusetts General Hospital (Other); Medical College of Wisconsin (Other); Medical University of South Carolina (Other); Hartford Hospital (Other)
Responsible Party: Principal Investigator, Magdy Selim, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2007P000288; 1R01NS057127-01A1 (NIH)
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Intracerebral Hemorrhage
Keywords: Deferoxamine; Safety; Intracerebral hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All participants will receive various dose-regimens of the study drug (deferoxamine mesylate). Each dose cohort will consist of at least 3 subjects.
  Interventions: Drug: Deferoxamine Mesylate

INTERVENTIONS:
Drug: Deferoxamine Mesylate — Various dose-regimens ranging from 7 mg/kg to 125 mg/kg (with a maximum allowable total daily dose of 6000 mg at any of the tested dose tiers, regardless of patient's weight), administered daily by IV infusion for three consecutive days.

SUMMARY:
Animal studies show that the breakdown of blood results in iron accumulation in the brain after brain hemorrhage (ICH); and that iron plays a role in brain injury in ICH patients. Deferoxamine (DFO) has been extensively used in clinical practice for more than 30 years to remove excessive iron from the body, and has been shown to provide some benefit in animal studies of ICH. Therefore, we plan to undertake this study to evaluate the safety and tolerability of treatment with DFO in patients with ICH, and to determine the maximal tolerated dose to be used in future studies to determine if treatment with DFO can improve the outcome of patients with ICH.

Our main objectives are: 1) to evaluate the safety and tolerability of varying doses of DFO, by determining the treatment related adverse events, in patients with ICH; and 2) to determine the maximal tolerated dose to be adopted in subsequent studies to test the efficacy of DFO in improving outcome after ICH.

We hypothesize that DFO is well-tolerated and has minimal serious adverse effects in patients with ICH; and that treatment with DFO will improve patients' outcome. The results can potentially bring into account new means to improve the outcome of patients with ICH. ICH is a frequent cause of disability and death. A successful study demonstrating the efficacy of iron-modifying therapy would be of considerable public health significance.

DETAILED DESCRIPTION:
An open-label, safety, tolerability, and dose-finding study using the continuous reassessment method.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. The diagnosis of ICH is confirmed by brain CT scan.
3. The first dose of the study drug can be administered within 18 hours of ICH symptom onset.
4. Signed and dated informed consent is obtained
5. Stable clinical and neurological status. Patients whose clinical or neurological status significantly deteriorates compared to presentation prior to administration of the study drug will be excluded.

Exclusion Criteria:

1. Previous chelation therapy or known hypersensitivity to DFO products
2. Abnormal renal function (serum creatinine > 2 mg/dl)
3. Known severe iron deficiency anemia
4. Planned surgical evacuation of ICH prior to administration of the study drug
5. Patients with suspected secondary ICH related to tumour, coagulopathy, ruptured aneurysm or arteriovenous malformation, or venous sinus thrombosis
6. Evidence of significant shift of midline brain structure (> 10 mm) or herniation on imaging studies.
7. Deep coma (Glasgow Coma Score (GCS) = 3-5) upon presentation
8. Taking iron supplements or prochlorperazine
9. Patients with heart failure taking > 500 mg of vitamin C daily
10. Known hearing impairment
11. Systolic blood pressure < 100 mmHg or diastolic blood pressure < 60 mmHg, confirmed by 3 consecutive readings
12. Significant chronic respiratory insufficiency
13. Known pregnancy (or positive pregnancy test), or breast-feeding
14. Patients known or suspected of not being able to comply with the study protocol due to alcoholism, drug dependency, incompliance, or any other cause.
15. Any condition which, in the judgement of the investigator, might increase the risk to the patient
16. Life expectancy of less than 90 days due to co-morbid conditions
17. Concurrent participation in another research protocol for investigation of another experimental therapy
18. Pre-existing Do Not Resuscitate (DNR) order, or indication that a new DNR order will be implemented within the first 48 hours of hospitalization. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities | First 7 days of hospitalization or diacharge, whichever occurs earlier

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Selim, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No